CLINICAL TRIAL: NCT07372417
Title: Role of Macrophage/Monocyte Mediated Inflammatory Response in Diminished Anesthetic Requirements During Aging
Brief Title: Macrophage/Monocyte Driven Inflammation and Anesthetic Sensitivity in Aging
Acronym: MACRO-AGE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC N°1538/25
Record Dates: First submitted 2025-11-17; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Aging; Inflammation; Blood-Brain Barrier Permeability; Anesthesia Brain Monitor; Anesthesia Depth Monitoring; Inflammation Biomarkers; Inflammaging; Monocyte
Keywords: Aging; Inflammation; General Anesthesia; Anesthetic Sensitivity; Cytokines; Alpha Oscillations; Blood Brain Barrier; Monocyte phenotype; macrophage phenotype
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples LCR samples if available Peritoneal lavage/biopsy if available
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults: Men and women requiring abdominal surgery aged 60 years or older.
- Young Adults: Men and women requiring abdominal surgery, aged 30 years or younger.

SUMMARY:
The goal of this observational study is to determine whether macrophage/monocyte mediated inflammatory signaling contributes to reduced anesthetic requirements in older adults undergoing major abdominal surgery. The main questions it aims to answer are:

* Is there a difference in anesthetic dosing requirements (minimum effective dose) between young and older patients undergoing major abdominal surgery?
* How do electroencephalographic (EEG) signatures under anesthesia correlate with age and systemic inflammatory markers?
* Is there an association between age, levels of circulating inflammatory cytokines, and monocyte/macrophage phenotypes with anesthetic requirements?

If there is a comparison group: Researchers will compare older adult patients undergoing major abdominal surgery to younger adult patients undergoing major abdominal surgery to see if macrophage/monocyte-mediated inflammatory signaling influences anesthetic sensitivity and the risk of postoperative neurocognitive complications in the older population.

Participants will:

* Receive general anesthesia for major abdominal surgery, with continuous recording of anesthetic dose requirements.
* Undergo electroencephalographic (EEG) monitoring during the anesthetic period.
* Provide blood samples for the measurement of circulating inflammatory cytokines and the assessment of monocyte phenotypes.
* Provide peritoneal tissue samples (collected during surgery) to evaluate tissue macrophage populations.
* Provide cerebrospinal fluid (CSF) samples to assess biomarkers of blood-brain barrier permeability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years or over 60 years old
* Scheduled for abdominal surgery
* General anesthesia planned with or without spinal anesthesia
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Chemotherapy or systemic corticosteroid use within the past 2 weeks.
* Pregnancy.
* Active sepsis or systemic infection.
* Emergency surgery.
* Requirement of ketamine or dexmedetomidine during the first hour of anesthesia.
* History or diagnosis of: stroke with persistent neurological deficit, dementia, Alzheimer's disease, Huntington's disease, amyotrophic lateral sclerosis, central nervous system autoimmune disorders, systemic autoimmune diseases, or infectious diseases of the central nervous system.
* Current treatment with immunomodulatory medications.
* Psychiatric disorders with psychotic features.
* Use of psychoactive or psychotropic recreational drugs within the week prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients from Hospital Clínico Universidad de Chile, in Santiago de Chile, that require elective abdominal surgery and are willing to participate in the study, meeting inclusion criteria and signing the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Frontal EEG alpha-band power | Perioperative
  Relative EEG alpha power during surgery under general anesthesia guided by standard age-adjusted dosing

SECONDARY OUTCOMES:
Time-to-loss of consciousness | Perioperative
  During propofol slow induction, the time required for unresponsiveness to verbal stimuli
Intraoperative anesthetic requirements | Perioperative
  Total dose and infusion rate of propofol and/or sevoflurane adjusted using frontal EEG monitoring
Time to emergence | Perioperative
  Time in minutes to eye opening since end of anesthesia, with verbal stimuli.
Cytokine circulating profile | Baseline
  Serum inflammatory cytokine profile
Monocyte/Macrophage phenotype in blood and peritoneal samples | Periprocedural
  inflammatory cell Pheontype present in circulating blood (monocytes) and in peritoneal lavage and tissue samples.
Blood-brain barrier permeability | Baseline
  CSF biomarkers present: albumin, cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Antonello Penna Silva, Anesthesia Professor, MD PhD, Study Chair — Brain and Anesthesia Laboratory (BAL), University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided